CLINICAL TRIAL: NCT06958822
Title: Estimation of the Incidence of Methemoglobinemia Associated With Ferric Carboxymaltose Administration
Brief Title: Ferric Carboxymaltose Methemoglobinemia Study
Acronym: FerMet
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Collaborators: Marmara University Pendik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Muhammet Özbilen, MD, Associate professor, Ordu University
Other Study IDs: 2024-KAEK-30 / 2025-43
Record Dates: First submitted 2025-04-13; First posted 2025-05-06 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-08

CONDITIONS: Methemoglobinemia; Anemia, Iron-Deficiency; Parenteral Iron Therapy; Ferric Carboxymaltose
Keywords: iron deficiency anemia; ferric carboxymaltose; intravenous iron; methemoglobinemia
MeSH Terms: conditions — Methemoglobinemia; Anemia, Iron-Deficiency | interventions — ferric carboxymaltose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- FCM Group: It will represent the group of patients who will be administered ferric carboxymaltose (FCM), i.e., the exposed group.
  Interventions: Drug: Ferric Carboxymaltose (FCM)
- Control Group: It will represent the control group of patients who do not receive FCM or any form of iron therapy, i.e., the unexposed group.

INTERVENTIONS:
Drug: Ferric Carboxymaltose (FCM) — As this is an observational study, ferric carboxymaltose recipients are determined based on routine medical care practices. The researchers do not define which participants will receive ferric carboxymaltose.
  Groups: FCM Group

SUMMARY:
Anemia that develops due to iron deficiency is called iron deficiency anemia. This common condition is treated with iron supplements taken either orally or given through an intravenous (IV) infusion. Ferric carboxymaltose (FCM) is one of the widely used, comparably newer IV iron preparations. Recently, several publications have raised the possibility that FCM may be associated with mild elevations in methemoglobin (metHb), a form of hemoglobin that cannot effectively deliver oxygen to tissues.

Methemoglobinemia is a known, though uncommon, side effect of some drugs. While usually mild and self-limiting, in certain cases it can become clinically significant or even life-threatening. This observational study is being conducted across multiple centers to better understand how often methemoglobinemia occurs after administration of FCM. As part of routine care, venous blood samples will be used to measure metHb levels in patients receiving FCM, and these results will be compared with those from individuals not exposed to the drug.

DETAILED DESCRIPTION:
Methemoglobinemia, which results from the conversion of ferrous iron (Fe2+) to ferric iron (Fe3+) in hemoglobin (Hb), is a potentially life-threatening disorder resulting in functional anemia due to reduced oxygen-carrying capacity. Methemoglobin (metHb) levels above one percent (>1%) are considered abnormal, and ≥3% metHb is considered clinically significant methemoglobinemia. Severe elevation of this level (>20%) leads to more dangerous clinical manifestations such as shortness of breath, confusion, arrhythmias, and seizures. Cases are usually asymptomatic until metHb levels reach 20%, and only discoloration of the blood and/or skin can be detected. Levels exceeding 70 percent are fatal.

The more common acquired form of methemoglobinemia, which can be congenital or acquired, is often caused by the use of drugs or toxic substances. Exposure to certain compounds that exceed the enzymatic reduction capacity of erythrocytes causes signs/symptoms. Benzocaine, phenazopyridine, dapsone, and nitrates/nitrites are the substances most commonly associated with methemoglobinemia.

Ferric carboxymaltose (FCM) is a third-generation intravenous iron drug with a ferric iron (Fe³⁺) compound that is widely used in the intravenous treatment of iron deficiency anemia. There are only three studies on the relationship between FCM and metHb reflected in the literature, one as a case report and two as congress proceedings. Given the expanding clinical use of FCM and the potential implications of undetected methemoglobinemia, there is a need to evaluate this association in a structured and systematic manner under routine care conditions. This study is designed to contribute to pharmacovigilance efforts by generating incidence data and exploring potential patient-related or treatment-related risk factors. Therefore, the investigators plan to determine the incidence of this comparably rare adverse effect with a prospective multicenter observational study.

The primary objective is to estimate the incidence of methemoglobinemia - defined as venous blood methemoglobin (metHb) levels ≥3%-within 30 min. following intravenous administration of ferric carboxymaltose in adult patients receiving routine care.

Secondary objectives include (i) description of the full distribution of metHb values post-infusion (ii) determination of whether metHb levels remain elevated beyond 30 min. in affected individuals, (iii) estimation of the background distribution of metHb levels in an unexposed, healthy outpatient population (iv) comparison of the metHb levels between FCM-exposed patients and unexposed controls (v) identification of potential associations between methemoglobinemia and relevant covariates, including patient demographics, total iron dose administered, baseline hemoglobin and venous oxygen saturation, or other potential oxidant exposures.

This study is a multicenter, prospective observational study. Ferric carboxymaltose recipients are determined based on routine medical care practices; the researchers do not define which participants will receive ferric carboxymaltose. Patient recruitment will take place between April 14, 2025, and September 15, 2025, per protocol, in 21 different health institutions.

Statistical analysis:

Methemoglobinemia rates (≥3% metHb) between the exposed (FCM) and unexposed groups will be compared using Fisher's exact test. Subgroup differences in continuous metHb levels will be analyzed using analysis of variance (ANOVA) with appropriate post hoc comparisons. Correlations between metHb levels and continuous clinical variables will be evaluated using correlation tests. Independent predictors of methemoglobinemia will be assessed through multivariable regression modeling. A two-sided significance threshold of α = 0.05 will be used for all tests.

ELIGIBILITY:
INCLUSION CRITERIA:

FCM Group:

1. Adults (≥18 years)
2. Presence of anemia (Hb <12 g/dl in women, <13 g/dl in men)
3. Low ferritin (<30 mcg/l)
4. Patients for whom FCM administration has been decided in routine medical care practice

Control Group:

Healthy adult (≥18 years) individuals who applied to the internal medicine outpatient clinic, who had no current or pre-existing chronic disease, who did not have anemia and iron deficiency (ferritin ≥30 mcg/L).

EXCLUSION CRITERIA:

1. Known methemoglobinemia-related diseases (Hb M disease, cytochrome b5 reductase deficiency, etc.)
2. Use of drugs associated with methemoglobinemia (acetylsalicylic acid, dapsone, chloroquine, metoclopramide, benzocaine, lidocaine, prilocaine, rasburicase, primaquine, sulfonamide, nitric oxide)
3. Those with B12 and/or folate deficiency
4. Those with Charlson Comorbidity Index ≥3
5. Presence of advanced organ failure (Stage 4 and 5 chronic kidney disease, Child C cirrhosis, NYHA class 3 and 4 chronic heart failure, respiratory failure requiring oxygen supplementation and similar processes)
6. Presence of malignancy (with or without cure)
7. Presence of active infection (CRP > 5 mg/dL) and/or other acute disorder/disease
8. Pregnancy status

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will consist of persons admitted to a total of 21 different secondary or tertiary care hospitals in 16 different provinces across Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 977 (Actual)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Clinically Significant Methemoglobinemia | From the time of enrollment through 30 minutes following completion of the infusion. If methemoglobin level is ≥3% after infusion, blood sampling will continue every half hour after the last blood gas for 24 hours until methemoglobinemia is <3%.
  Methemoglobin levels will be measured just before the infusion and at the 15th and 30th minutes post-infusion through venous sampling. The levels equal to or above 3% will be regarded as clinically significant methemoglobinemia.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet Özbilen, MD, Study Director — Ordu University Faculty of Medicine; Gökhan Tazegül, MD, Study Director — Marmara University; Volkan Aydın, MD PhD, Study Director — Marmara University School of Dentistry; Murat Bahadır, MD, Principal Investigator — Ordu University Faculty of Medicine, Department of Internal Medicine; Bilge Ada Özcan, MD, Principal Investigator — Marmara University Training and Research Hospital; Mehmet Bankir, MD, Principal Investigator — University of Health Sciences Adana City Health Application and Research Center; Mehmet Can Erişen, MD, Principal Investigator — University of Health Sciences Adana City Health Application and Research Center; Nurhayat Özkan Sevencan, MD, Principal Investigator — Karabuk University Training and Research Hospital; Ceren Çevik, MD, Principal Investigator — Karabuk University Training and Research Hospital; Aysel Toçoğlu, MD, Principal Investigator — Sakarya University Training and Research Hospital; Sümeyye Çekiç, MD, Principal Investigator — Sakarya University Training and Research Hospital; Arzu Denler Kılıç, MD, Principal Investigator — Çankırı State Hospital; Mehmet Selim Mamiş, MD, Principal Investigator — Siirt University Faculty of Medicine Training and Research Hospital; Necip Nas, MD, Principal Investigator — Siirt University Faculty of Medicine Training and Research Hospital; Teslime Ayaz, MD, Principal Investigator — Izmir Bakircay University Cigli Training and Research Hospital; Barış Emekdaş, MD, Principal Investigator — Izmir Bakircay University Cigli Training and Research Hospital; İhsan Solmaz, MD, Principal Investigator — University of Health Sciences Diyarbakır Gazi Yaşargil Training and Research Hospital; Ömer Faruk Alakuş, MD, Principal Investigator — University of Health Sciences Diyarbakır Gazi Yaşargil Training and Research Hospital; Kamil Konur, MD, Principal Investigator — Recep Tayyip Erdoğan University Faculty of Medicine Training and Research Hospital; Hasan Sözel, MD, Principal Investigator — Akdeniz University Hospital; Esin Avşar Küçükkurt, MD, Principal Investigator — Akdeniz University Hospital; Hacer Şen, MD, Principal Investigator — Balıkesir University Health Practice and Research Hospital; Özge Kama Başçı, MD, Principal Investigator — Balıkesir University Health Practice and Research Hospital; Nizameddin Koca, MD, Principal Investigator — Bursa City Hospital; Fatih İleri, MD, Principal Investigator — Bursa City Hospital; Banu Açmaz, MD, Principal Investigator — Kayseri City Hospital; Erdem Aydın, MD, Principal Investigator — Kayseri City Hospital; İdris Baydar, MD, Principal Investigator — Mardin Artuklu University Training and Research Hospital; Şengül Baran Yerlikaya, MD, Principal Investigator — Mardin Artuklu University Training and Research Hospital; Yıldız Okuturlar, MD, Principal Investigator — Mehmet Yılmaz Aydınlar Acıbadem University; Sibel Serin Ocak, MD, Principal Investigator — Umraniye Training and Research Hospita; Nur Düzen Oflas, MD, Principal Investigator — Van Yüzüncü Yıl University Training and Research Hospital; Abdullah Güneş, MD, Principal Investigator — Van Yüzüncü Yıl University Training and Research Hospital; Nazire Osmançelebioğlu, MD, Principal Investigator — Recep Tayyip Erdoğan University Faculty of Medicine Training and Research Hospital; Ant Uzay, MD, Principal Investigator — Mehmet Yılmaz Aydınlar Acıbadem University; Sevgi Gülşen Koç, MD, Principal Investigator — Antalya City Hospital; Ayşe Karaduru, MD, Principal Investigator — Antalya City Hospital; Gamze Kocaman, MD, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital; Ali Erol, MD, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital; Mehmet Biricik, MD, Principal Investigator — Mardin Kiziltepe State Hospital; Emine Binnetoğlu, MD, Principal Investigator — Çorlu Vatan Hospital; Muhammet Fatih Şahin, MD, Principal Investigator — Bursa Kestel State Hospital; Ebru Çağrı Çakır Özden, MD, Principal Investigator — Bursa Kestel State Hospital
Locations (23):
- Turkey (Türkiye) (23):
  - University of Health Sciences Adana City Health Application and Research Center, Adana, Adana
  - Akdeniz University Hospital, Konyaalti, Antalya
  - Balıkesir University Health Practice and Research Hospital, Merkez, Balıkesir
  - Bursa City Hospital, Nilufer, Bursa
  - University of Health Sciences Diyarbakır Gazi Yaşargil Training and Research Hospital, Kayapınar, Diyarbakır
  - Mehmet Yılmaz Aydınlar Acıbadem University, Ataşehir, Istanbul
  - Marmara University Training and Research Hospital, Pendik, Istanbul
  - Umraniye Training and Research Hospital, Ümraniye, Istanbul
  - Izmir Bakircay University Cigli Training and Research Hospital, Çiğli, İzmir
  - Karabuk University Training and Research Hospital, Karabük, Karabük Province
  - Kayseri City Hospital, Kocasinan, Kayseri
  - Antalya City Hospital, Antalya, Kepez
  - Bursa Kestel State Hospital, Bursa, Kestel
  - Mardin Kızıltepe State Hospital, Mardin, Kızıltepe
  - Mardin Artuklu University Training and Research Hospital, Merkez, Mardin
  - Ordu University Training and Research Hospital, Altinordu, Ordu
  - Recep Tayyip Erdoğan University Faculty of Medicine Training and Research Hospital, Rize, Rize Province
  - Sakarya University Training and Research Hospital, Adapazarı, Sakarya
  - Siirt University Faculty of Medicine Training and Research Hospital, Siirt, Siirt
  - Van Yüzüncü Yıl University Training and Research Hospital, Merkez, Van
  - Bursa Yuksek Ihtisas Training and Research, Bursa, Yıldırım
  - Çankırı State Hospital, Çankırı, Çankırı
  - Çorlu Vatan Hospital, Tekirdağ, Çorlu

IPD SHARING:
Plan to Share IPD: Yes
Age, gender, hemoglobin, MCV, MCHC, ferritin, CRP, transferrin saturation, ferric carboxymaltose (FCM) drug dose, FCM infusion concentration, infusion duration, methemoglobin levels
Supporting Information: Study Protocol
Time Frame: Beginning 3 months after publication with no end date
Access Criteria: De-identified individual participant data (IPD) that underlie the results reported in this article (text, tables, figures, and appendices) will be made available to researchers who provide a methodologically sound proposal in order to achieve aims in the approved proposal.
  Access to the IPD will require prior approval from the principal investigator. Researchers will need to submit a formal data access request including:
  A detailed research protocol with clear objectives and statistical analysis plan,
  A data use agreement,
  Proof of institutional ethics approval (if applicable).
  Decisions regarding data access will be made by the study's data sharing committee within a reasonable time frame, and applicants will be notified via email.
  Requests should be directed to: drozbilen@gmail.com
  Data will be shared via a secure data transfer system or repository, depending on the nature and size of the dataset.

REFERENCES:
- [Background] Tazegul Gokhan, Kimyon Yusuf, Odabasi Zekaver. Ferric carboxymaltose induced methaemoglobinemia: Preliminary data of a novel side effect. 22nd European Congress of Internal Medicine , İstanbul, Turkey, 2024.
- [Background] Özbilen M, Savrun ŞT, Aygün A, Kaya Y. P1492: A New Potential And Prevalent Side Effect of Ferric Carboxymaltose: Methemoglobinemia. A Case-Control Study. Hemasphere. 2023 Aug 8;7(Suppl 3):e825173f.
- [Background] Ozbilen M, Savrun ST, Aygun A, Kaya Y. Ferric Carboxymaltose-mediated Methemoglobinemia. Curr Drug Saf. 2024;19(1):134-137. doi: 10.2174/1574886318666230213111038. PMID 36779493